CLINICAL TRIAL: NCT06549933
Title: The Influence of Cryostimulation on Reducing Inflammation and Improving Motor Skills in Football Player
Brief Title: The Effect of Cryostimulation on Inflammation and Motor Functions. The Study Was Conducted to Determine the Effect of Five Days of Whole-body Cryostimulation (PBC) on Reducing Inflammation and Improving Motor Skills in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Kriokomora 845/22; 12622001541796 (Registry Identifier: ANZCTR of Australia and New Zealand)
Record Dates: First submitted 2024-07-24; First posted 2024-08-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-07

CONDITIONS: Rest; Training
Keywords: cryostimulation; regeneration; football players; inflammation; motor functions
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Athletes undergoing regular training were divided into two groups. One of them was subjected to cryotherapy treatments, the other was a control group, not subjected to any treatments at that time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cryostimulation (Experimental): Cryostimulation performed in a cryosauna for five consecutive days.
  Interventions: Other: Criostymulation

INTERVENTIONS:
Other: Criostymulation — Method: Cryosauna. Temperature: -160°C. Duration: 5 days. Session Timing: 9:00 a.m.
  Session Length: 3 minutes per day

SUMMARY:
The aim of the study was to determine the effect of a 5-day PBC on reducing inflammation and improving motor skills in soccer players during the initial phase of the training period.

The five-day cryostimulation applied did not significantly affect the profile of inflammatory markers in soccer players. However, a reduction in visuo-motor reaction time (RT) was registered in PBC-treated soccer players, suggesting the potential benefits of this method in improving motor skills.

DETAILED DESCRIPTION:
Cryostimulation is one of the methods of post-exercise recovery, involving short-term (3 min) exposure of the body to extremely low temperatures, oscillating between -100°C and -190°C. The purpose of this therapy is to reduce inflammation, reduce physical and mental fatigue and use it as a passive form of preparing the body for further exercise as part of the training process.

The study was conducted to determine the effect of five days of whole-body cryostimulation (PBC) on reducing inflammation and improving motor skills in soccer players. A group of 24 football players was randomly divided into a test group (PBC; -140°C ± 20°C, 3 min, 5 days) and a control group (CON). Before the cryostimulation session, both groups were subjected to visual-motor ability tests, which were repeated on the last day of the study. Blood samples were collected at four time points (P0-1 day, P1-3 day, P2-5 day, P3-2 days after the test). Levels of creatine kinase (CK), tumor necrosis factor (TNFα), interleukins (IL-6, IL-10), testosterone (T) and cortisol (C) were determined in the samples.

ELIGIBILITY:
Inclusion Criteria:

* athletes
* no previous experience with systemic cryotherapy
* any other forms of recovery or cosmetic treatments

Exclusion Criteria:

* alcohol or any other stimulants
* anti-inflammation drugs
* injuries

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-02-24 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
IL-6 (Interleukin-6) | Before, after 3 days and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit
TNF-alpha (Tumor necrosis factor-alpha) | Before, after 3 days and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit
IL-10 (Interleukin-10) | Before, after 3, and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit
CK (creatine kinase) | Before, after 3, and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit
Cortisol | Before, after 3, and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit
Testosterone | Before, after 3, and 5 days of cryostimulation
  Immunoenzymatic assay method using a diagnostic ELISA Kit

SECONDARY OUTCOMES:
Anthropometric measurments | Before, after 3, and 5 days of cryostimulation
  Analysis of body composition, Tanita BC-418

CONTACTS AND LOCATIONS:
Overall Officials: Izabela Różycka, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No